CLINICAL TRIAL: NCT04208737
Title: Comparing Effects of Recruitment Maneuver on Functional Residual Capacity in Patients Undergo Laparoscopic Surgery : A Randomized Prospective Study.
Brief Title: Effects of Recruitment Maneuver on Functional Residual Capacity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Nuzhet Mert Senturk, MD, Prof, Prof.Dr., Istanbul University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2018/938
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Anesthesia; Surgery; Atelectasis
MeSH Terms: conditions — Pulmonary Atelectasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): 3 FRC measurements will be perforemed, whereby : First measurement; after aneshesia induction and intubation. Second measurement; after pneumoperitoneum Third measurement; end of the operation
  After the operation,Postoperative Room Air Test (RAT) will be applied.
- study group (Experimental): 5 FRC measurements will be performed We will apply recruitment maneuver two times to patients with 30cmH2O pressure for 15 seconds .
  First Recruitment maneuver will be applied after the fşrst measurement of FRC following intubation Second Recuitment maneuver will be applied at the end of operation
  First FRC measurement after anesthesia induction and intubation. Second FRC measurement after first recruitment maneuver Third FRC measurement; after pneumoperitoneum Fourth FRC measurement before second recruitment maneuver Fifth FRC measurement after second recruitment maneuver and at the end of operation
  Interventions: Procedure: recruitment maneuver

INTERVENTIONS:
Procedure: recruitment maneuver — 30 cmH2O pressure 15 seconds
  Arms: study group

SUMMARY:
Recruitment maneuver is frequently used in daily anaesthesia routine to prevent athelectasia and ventilation perfusion mismatch. Especially pneumoperitoneum in laparoscopic surgeries affects the functional residual capacity (FRC) negatively. Recently, FRC can be measured at bedside in intensive care units.

The lack of studies evaluating FRC measurements peroperatively and how recruitment maneuvers affect it, attract attention.

DETAILED DESCRIPTION:
An ICU-ventilator capable to measure the FRC will be used for the mechanical ventilation in patients undergıoing laparoscopic surgery, where anaesthesia maintenance will be achieved with TIVA.

FRC will be measured in different steps of the operation. In the study group, a recruitment manover will be applied to evaluate its effects on FRC.

ELIGIBILITY:
Inclusion Criteria:

1-18-65 years age 2-no lung disease 3-laparoscopic cholecystectomies surgery

Exclusion Criteria:

1. <18 years old
2. >65 years old
3. denial of patient
4. patients having one of: lung disease, cardiac failure, severe cardiac valvular disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-12-23 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Comparison of FRC measurements at beginning and end of anesthesia | within max 5 minutes after the intubation and with max 5 minutes before the extubation
  First FRC will be measured after ; the last FRC will be measure bedore the extubation

SECONDARY OUTCOMES:
Positive room air test | in recovery room 30 minutes after operation
  in recovery room when patient modified aldrete score ≥ 9 patient SPO2 when breathing in room air If patients' spo2 value ≤ 96%, named as room air test positive

CONTACTS AND LOCATIONS:
Overall Officials: Elif Aygun, MD, Principal Investigator — Istanbul University
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul University, Istanbul
  - Istanbul University, Department of Anesthesiology, Istanbul

IPD SHARING:
Plan to Share IPD: No